CLINICAL TRIAL: NCT02352389
Title: A Pilot Study of Influenza Viruses Isolated From Immunocompromised Children and Adolescents
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FLUMUT
Record Dates: First submitted 2015-01-22; First posted 2015-02-02 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Influenza, Human
Keywords: Childhood; Cancer; Genetic mutations
MeSH Terms: conditions — Influenza, Human; Neoplasms | interventions — Blood Specimen Collection; Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Influenza: Children and young adults identified as having influenza infections by the St. Jude Children's Research Hospital diagnostic microbiology will be approached to participate in the study. Biological samples will be collected on Day 0 within 72 hours of the diagnosis of influenza, and at 7, 14, 21, and 28 days later.
  Interventions: Symptom checklist, Blood sample, Nasal swab, Oropharyngeal swab, Stool sample.
  Interventions: Other: Blood sample; Other: Nasal swab; Other: Oropharyngeal swab; Other: Stool sample; Other: Symptom checklist

INTERVENTIONS:
Other: Blood sample — Blood samples will be drawn and analyzed at Day 0, 7, 14, 21, and 28
  Other Names: Blood work
Other: Nasal swab — Obtained on Day 0, 7, 14, 21 and 28.
  Other Names: Mid-turbinate swab
Other: Oropharyngeal swab — Obtained on Day 0, 7, 14, 21 and 28.
  Other Names: Throat swab
Other: Stool sample — Obtained on Day 0, 7, 14, 21 and 28.
  Other Names: Stool specimen
Other: Symptom checklist — Obtained on Day 0, 7, 14, 21 and 28.
  Other Names: History

SUMMARY:
The purpose of the proposed study is to gather critical information that may be useful in designing effective prevention and treatment strategies for control of seasonal influenza and an influenza pandemic. In particular, the critical questions are related to the virus' ability to adapt to efficient replication and spread in humans.

Influenza is a contagious respiratory illness caused by influenza A and B viruses. Influenza infections result in about 230,000 hospitalizations and 36,000 deaths annually in the United States. Children with cancer are more likely to have serious influenza and complications than those who have no underlying medical problems. They are also more likely to have prolonged influenza illnesses and to shed influenza viruses from their noses for long periods of time (sometimes for months). Recent studies suggest that influenza viruses may also be carried and shed from the gastrointestinal tract. New types of influenza viruses emerge frequently through mutations that occur when the viruses replicate. These mutations allow the virus to escape from killing by the immune system and are, in large part, responsible for seasonal epidemics of influenza that occur in the fall or winter months. It is possible that viruses can mutate when they are carried in the respiratory or gastrointestinal tracts for long periods, potentially giving rise to viruses that spread more easily to other persons, cause more severe disease, lead to new influenza epidemics or make the viruses resistant to drugs used to treat influenza.

Researchers at St. Jude Children's Research Hospital want to learn about how influenza viruses mutate in immunocompromised children. They will investigate how long children with cancer carry influenza viruses in their nose, throat and gastrointestinal tract and the characteristics of any mutations that are found in these viruses.

DETAILED DESCRIPTION:
Participants will have nasal, oral and stool specimens obtained at the time they are diagnosed with influenza infections, and 7, 14, 21 and 28 days later. The genome of influenza viruses that are isolated from these participants will be sequenced and compared to one another and to standard influenza strains.

PRIMARY OBJECTIVE:

* To determine the proportion of pediatric oncology patients with nasal and oropharyngeal shedding of influenza viruses at 7, 14, 21 and 28 days following the diagnosis of infection.

SECONDARY OBJECTIVES:

* To determine the proportion of gastrointestinal shedding of human influenza viruses.
* To determine the frequency and pattern of mutations in influenza viruses isolated from pediatric oncology patients.
* To explore the biological consequences of mutations in influenza viruses isolated from pediatric oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Less than 22 years of age.
* Currently receiving active therapy for malignant disease at St. Jude, excepting surgical therapy only, or has received a hematopoietic stem cell transplant in the last 6 months.
* Subject has had a positive test for influenza (by direct fluorescent antibody, nucleic acid amplification test or viral culture) within 72 hrs of the time of enrollment.
* Agrees to participate in the study.
* Able to understand and comply with planned study procedures.
* Is available for all study visits.

Exclusion Criteria:

* Contraindication to nasal (mid-turbinate) swabs (e.g. nasal lesion or obstruction)
* Has any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Previous enrollment on study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults identified as having influenza infections by the St. Jude Children's Research Hospital diagnostic microbiology will be approached to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with nasal shedding of influenza viruses | Day 0
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with nasal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with nasal shedding of influenza viruses | Day 7
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with nasal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with nasal shedding of influenza viruses | Day 14
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with nasal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with nasal shedding of influenza viruses | Day 21
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with nasal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with nasal shedding of influenza viruses | Day 28
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with nasal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with oropharyngeal shedding of influenza viruses | Day 0
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with oropharyngeal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with oropharyngeal shedding of influenza viruses | Day 7
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with oropharyngeal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with oropharyngeal shedding of influenza viruses | Day 14
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with oropharyngeal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with oropharyngeal shedding of influenza viruses | Day 21
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with oropharyngeal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Proportion of patients with oropharyngeal shedding of influenza viruses | Day 28
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of pediatric oncology patients with oropharyngeal shedding of influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.

SECONDARY OUTCOMES:
Frequency of gastrointestinal shedding of human influenza virus | Day 0
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of gastrointestinal shedding of human influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided. Frequency of gastrointestinal shedding of human influenza virus and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of gastrointestinal shedding of human influenza virus | Day 7
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of gastrointestinal shedding of human influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided. Frequency of gastrointestinal shedding of human influenza virus and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of gastrointestinal shedding of human influenza virus | Day 14
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of gastrointestinal shedding of human influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided. Frequency of gastrointestinal shedding of human influenza virus and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of gastrointestinal shedding of human influenza virus | Day 21
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of gastrointestinal shedding of human influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided. Frequency of gastrointestinal shedding of human influenza virus and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of gastrointestinal shedding of human influenza virus | Day 28
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of gastrointestinal shedding of human influenza viruses and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided. Frequency of gastrointestinal shedding of human influenza virus and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of mutations in influenza viruses | Day 0
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of human influenza viruses with mutations and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of mutations in influenza viruses | Day 7
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of human influenza viruses with mutations and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of mutations in influenza viruses | Day 14
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of human influenza viruses with mutations and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of mutations in influenza viruses | Day 21
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of human influenza viruses with mutations and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Frequency of mutations in influenza viruses | Day 28
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as proportion of human influenza viruses with mutations and its 95% confidence interval at days 7, 14, 21, and 28 days will be provided.
Number of mutations by type in influenza viruses | Day 0
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the type of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days will be provided to show the pattern of mutations. Genetic variants are defined to meet a minimum minor allele frequency of 20%.
Number of mutations by type in influenza viruses | Day 7
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the type of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days will be provided to show the pattern of mutations. Genetic variants are defined to meet a minimum minor allele frequency of 20%.
Number of mutations by type in influenza viruses | Day 14
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the type of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days will be provided to show the pattern of mutations. Genetic variants are defined to meet a minimum minor allele frequency of 20%.
Number of mutations by type in influenza viruses | Day 21
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the type of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days will be provided to show the pattern of mutations. Genetic variants are defined to meet a minimum minor allele frequency of 20%.
Number of mutations by type in influenza viruses | Day 28
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the type of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days will be provided to show the pattern of mutations. Genetic variants are defined to meet a minimum minor allele frequency of 20%.
Biological consequences of mutations in influenza viruses | Day 0
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days that are associated with antiviral resistance will be provided to show the biological consequences. Two-sample t-tests or Wilcoxon rank-sum tests will be performed as appropriate to compare isolates to parental influenza isolates from the same patients.
Proportion of mutations in influenza viruses by collection site | Day 7
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days that are associated with antiviral resistance will be provided to show the biological consequences. Two-sample t-tests or Wilcoxon rank-sum tests will be performed as appropriate to compare isolates to parental influenza isolates from the same patients.
Proportion of mutations in influenza viruses by collection site | Day 14
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days that are associated with antiviral resistance will be provided to show the biological consequences. Two-sample t-tests or Wilcoxon rank-sum tests will be performed as appropriate to compare isolates to parental influenza isolates from the same patients.
Proportion of mutations in influenza viruses by collection site | Day 21
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days that are associated with antiviral resistance will be provided to show the biological consequences. Two-sample t-tests or Wilcoxon rank-sum tests will be performed as appropriate to compare isolates to parental influenza isolates from the same patients.
Proportion of mutations in influenza viruses by collection site | Day 28
  Day 0 is collected within 72 hours of diagnosis of influenza. Descriptive statistics, such as the proportion of mutations observed in human influenza viruses at days 7, 14, 21, and 28 days that are associated with antiviral resistance will be provided to show the biological consequences. Two-sample t-tests or Wilcoxon rank-sum tests will be performed as appropriate to compare isolates to parental influenza isolates from the same patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth E. Adderson, MD, MSc, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols